CLINICAL TRIAL: NCT02446002
Title: Assessment of the Effect of Naltrexone on Lofexidine Single Dose Pharmacokinetics in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM-LX1-1009; 1R01DA030916 (Other Grant/Funding Number: National Institute on Drug Abuse)
Record Dates: First submitted 2015-05-07; First posted 2015-05-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Volunteer
MeSH Terms: interventions — lofexidine; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lofexidine + Naltrexone (Experimental)
  Interventions: Drug: Lofexidine + Naltrexone

INTERVENTIONS:
Drug: Lofexidine + Naltrexone — Lofexidine HCl (two 0.2 mg tablets) will be administered as a single oral dose (0.4 mg) on Day 1 and on Day 11.Commercially available naltrexone HCL tablets will be administered as a single oral 25 mg dose on Day 4 and as a single oral 50 mg dose on Days 5 through 13. On Day 11 administration of both naltrexone and lofexidine will occur. Dose administration times for each drug are to be standardized for all treatment days. The scheduling of the naltrexone dose is to be standardized so that the naltrexone dose is administered 2 hours after the lofexidine dose on Day 11 when both drugs are administered.
  Other Names: Lofexidine HCL; Naltrexone HCL

SUMMARY:
A Phase 1, open-label, single-arm study with two single doses of lofexidine and multiple doses of naltrexone in healthy adult subjects to determine the effect of naltrexone on the single dose pharmacokinetics of the oral lofexidine formulation.

DETAILED DESCRIPTION:
Subjects will be confined to an inpatient facility for a total of 14 nights and 15 days. Subjects who successfully complete screening will report to the inpatient facility (Day -1). At Day 1 all subjects will receive the first single, oral dose of 0.4 mg lofexidine HCl (two 0.2 mg tablets) dosed with 240 mL of water (no food). The lofexidine dose will be followed by a 74-hour interval before beginning naltrexone daily dosing on Day 4 .The first naltrexone administration on Day 4 will be at a dose of approximately 25 mg QD, with subsequent doses on Days 5 to 13 at 50 mg QD. On Day 11, the second single dose of lofexidine (0.4 mg) will be administered and followed by the daily administration of the naltrexone dose (50 mg). The daily administration of naltrexone dose (50 mg) will continue on Day 12 and Day 13.After each administration of lofexidine on Day 1 and Day 11, fingerstick blood samples will be collected for lofexidine pharmacokinetic (PK) analysis before dosing and after dosing at multiple time points.Safety will be assessed by recording adverse events (AEs), measuring vital signs (blood pressure and pulse rate) and clinical laboratory tests (chemistry, hematology, and urinalysis), recording 12-lead safety and Holter electrocardiograms (ECGs), and performing physical exams.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 35 kg/m^2
* females of childbearing potential must be using contraception or must be surgically sterile
* Subject is in good health based on medical history, physical exam, laboratory profile, electrocardiogram (ECG) as judged by investigator
* If subject smokes, subject agrees to limit smoking while in the study to not more than 10 cigarettes per day
* Subject provides written informed consent before participation in the study, and an appropriate HIPAA (Health Insurance Portability and Accountability Act) form is signed and dated

Exclusion Criteria:

* Subject has a history of clinically significant disease, including cardiovascular, gastrointestinal (GI), renal, hepatic, pulmonary, endocrine, hematologic, vascular, immunologic, metabolic, or collagen disease.
* Females: pregnant, breastfeeding, planning to become pregnant, or a positive pregnancy test.
* Clinically significant illness within 4 weeks before Day -1.
* Use of herbal supplements within 3 weeks before Day -1.
* Received treatment of more than a single dose of a CYP3A4 inducer (e.g., rifampin, barbiturates, phenytoin, glucocorticoids, St. John's Wort) within 4 weeks before Day -1.
* Received treatment with a strong CYP3A4 inhibitor (e.g., ketoconazole, diltiazem, macrolide antibiotics) within 2 weeks before Day -1.
* Currently taking any medication identified as potentially producing QTc prolongations of 10 msec or greater.
* Received an investigational medication during the last month (30 days) preceding Day -1.
* Consumes more than 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) or has a significant history of alcohol abuse or drug/chemical abuse within the last 1 year.
* Consumed grapefruit, grapefruit juice, Seville oranges, and/or starfruit within 4 days before Day -1.
* Positive urine drug or alcohol screen, unless positive result is due to an approved prescribed medication (e.g., pain medication or benzodiazepine).
* Positive human immunodeficiency virus (HIV) test or tests positive for hepatitis B surface antigen.
* Known allergy or intolerance to any compound in the test product or any other closely related compound.
* Donated blood/plasma, exceeding 500 mL, during the 3-month period before Day -1.
* Abnormal cardiovascular exam at Screening, including any of the following: clinically significant abnormal ECG (e.g., second or third degree heart block, uncontrolled arrhythmia, QTcF [Fridericia's correction] interval >450 msec for males and >470 msec for females); pulse<45 bpm or symptomatic bradycardia; systolic blood pressure <90 mmHg or symptomatic hypotension; blood pressure >165/95 mmHg; or prior history of myocardial infarction within 1 year before Day -1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
PK Profile for Lofexidine only: Cmax, Tmax, AUC, AUC 0-24, AUC 0-t, AUC 0-infinity, λz, and CL/F | Day 1 through Day 11
  Descriptive statistics will be used to summarize lofexidine concentrations at each time point and PK parameters by treatment phase.Comparisons will be made between Day 1 and Day 11 for Cmax, AUC0-24, AUC0-t, AUC0-∞, Tmax, and t1/2
PK Profile for Naltrexone only: Cmax, AUC0-24, Tmax, and CL/F | Day 4 through Day 11
  Descriptive statistics will be used to summarize naltrexone concentrations at each time point and PK parameters by treatment phase. Comparisons will be made between Day 10 and Day 11 for Cmax, AUC0-24, and Tmax at steady-state.

SECONDARY OUTCOMES:
All Adverse Events (AEs) and Serious Adverse Events (SAEs) will be reported throughout the study and will include all subjects who receive at least 1 dose of study medication. | Day 1 through 14
  Treatment phases include lofexidine alone/washout [Days 1-3]; naltrexone alone [Days 4-10]; and lofexidine plus naltrexone [Days 11-14]

CONTACTS AND LOCATIONS:
Overall Officials: George Atiee, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States